CLINICAL TRIAL: NCT00846222
Title: Adjunctive Mild Hypothermia Therapy to Primary Percutaneous Coronary Intervention in Patients With Acute Myocardial Infarction Complicated With Shock: A Feasibility Study
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Responsible Party: Alex Blatt MD, Assaf Harofeh MC
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192/08
Record Dates: First submitted 2009-02-16; First posted 2009-02-18 (Estimated); Last update posted 2009-02-18 (Estimated); Status verified 2009-02

CONDITIONS: Myocardial Infarction Complicated With Cardiogenic Shock

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mild theraputic hypothermia (Experimental)
  Interventions: Procedure: Hypothermia

INTERVENTIONS:
Procedure: Hypothermia — Mild therapeutic hypothermia, 33-34 celsius, for 12 hours

SUMMARY:
The purpose of this study is evaluate the safety and feasibility of mild therapeutic hypothermia (TH) during and 12 hours after primary percutaneous coronary intervention for acute myocardial infarction complicated with shock

ELIGIBILITY:
Inclusion Criteria:

* Recent myocardial infarction: 24 hours of start pain
* Pump failure cardiogenic shock (defined as persistent hypotension, systolic BP < 90 mmHg, despite fluids and catecholamines infusion, with tissue hypoperfusion signs
* Candidate for immediate percutaneous reperfusion
* Maximal care support: mechanical ventilation, intraaortic balloon contrapulsation

Exclusion Criteria:

* Cardiogenic shock related to mechanical complication: free wall rupture, acute mitral regurgitation, acute VSD, tamponade
* Pregnant women
* Absence of maximal support care

Ages: 18 Years to 88 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2009-02; Primary Completion 2010-04 (Estimated); Study Completion 2010-07 (Estimated)

PRIMARY OUTCOMES:
Primary en point: presence of major adverse cardiac events (MACE) MACE definition: death and non-fatal re-infarction. | 30 days

SECONDARY OUTCOMES:
Infarct size calculated by area under thr curve creatinine kinase according consecutive samples Reversal stunning by blinded observer echocardiographic assessment | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf Harofeh MC, Ẕerifin, Israel

REFERENCES:
- [Background] Dixon SR, Whitbourn RJ, Dae MW, Grube E, Sherman W, Schaer GL, Jenkins JS, Baim DS, Gibbons RJ, Kuntz RE, Popma JJ, Nguyen TT, O'Neill WW. Induction of mild systemic hypothermia with endovascular cooling during primary percutaneous coronary intervention for acute myocardial infarction. J Am Coll Cardiol. 2002 Dec 4;40(11):1928-34. doi: 10.1016/s0735-1097(02)02567-6. PMID 12475451
- [Background] Hale SL, Dave RH, Kloner RA. Regional hypothermia reduces myocardial necrosis even when instituted after the onset of ischemia. Basic Res Cardiol. 1997 Oct;92(5):351-7. doi: 10.1007/BF00788947. PMID 9486356